CLINICAL TRIAL: NCT04892927
Title: NCI SBIR Contract for Patient Navigation Tool Prototype Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GMG Arcdata LLC (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: 75N91020C00043; 75N91020C00043-0-9999-1 (NIH)
Record Dates: First submitted 2021-05-02; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Pancreas Cancer; Hepatobiliary Cancer; Patient Engagement
MeSH Terms: conditions — Pancreatic Neoplasms; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
GMG ArcData will create a mobile-based application to improve communications and data exchange among patients and navigators involved in new pancreas surgery oncology episodes of care. Functionality will align with care processes using smartphone and the EHR patient portal. GMG will apply user-centered design theory and behavioral psychology approaches to co-design, develop, and test usability of features that optimize patient navigators-patient encounters on scheduling issues, nutrition guidance, pain management, wellbeing assessments, and activity tracking. Evaluation endpoints will reflect how the application improves the efficiency of workflows and lessens cognitive burden. Study will assess how patients and navigators perceive the tool's ability to provide more control and easier access to information about surgical care. The key project innovations are based on Fast Healthcare Interoperability Resources (FHIR)-based engineering standards that enable interoperability among digital health platforms, apply 'recommender' functions based on similar patients' experiences, and exploit microeducation tools to enhance patient understanding about their surgical care. The research team has partnered with MedStar Health and Georgetown University Lombardi Comprehensive Cancer Center to co-design the software and access patients for usability testing. Successful implementation will lead to exploring a joint venture for scaling to other care episodes, expanded functionality, and co-creating business models for commercialization.

DETAILED DESCRIPTION:
The objective of this Phase I Small Business Innovation Research project is to determine the scientific or technical feasibility of R&D efforts. The requirements that will be addressed include:

1. Reducing the cognitive or time burden (or both) of navigation-related tasks performed by either patient navigators (PNs) or patients;
2. Integrating seamlessly into the workflow of PNs and existing health information technology (IT) architecture; and
3. Transmitting information securely across a variety of IT systems.

The study's proposed approach for developing software to support pancreatic cancer patient navigation across the care continuum will be addressed through research addressing these three Specific Aims:

1. Engineering concepts that embrace interoperability through leveraging open messaging standards and improve usability by adopting human-centered design principles at project inception. With respect to interoperability, the key facet of this work's innovation will be using interoperability standards (e.g., FHIR) to interface with an electronic health record (EHR) at an NCI-designated Comprehensive Cancer Center. Doing so will facilitate scalability and flexibility in functionality that enhances the user experience for integrated functions (patient care information delivery, patient assessment, pain assessment, nutrition and activity). The study will apply user-centered design features that will allow us to assess patient engagement, efficiency of information flow, and navigator satisfaction.
2. Research, design, and potential implementation of open source solutions for recommender systems. Smart recommendations, nudges, and automation enable users, both patients and PNs, to receive certain actionable options for an interaction based on experiences from other patients and navigators with similar preferences or share similar characteristics. The adoption of this approach will address cognitive overload, diminish presentation of unnecessary or inapplicable content, and create enhanced user experiences and more efficient and effective decision making.
3. Research, design, and potential implementation of enhanced content delivery using asynchronous microeducation features. The most common approach to patient education is to create flat files or pdfs that are shared with patients for instruction. The study plans to demonstrate the value of instructional design in the software application to enhance patient engagement and understanding. Video features of the patient experience can be enhanced with videography, 360 immersive videos (for instance to show the patient the inside of the operating and recovery rooms). Through these delivery platforms content can be evaluated with AB testing to assess patient's responsiveness (for example, wound care, graphic representation of the anatomical surgical approach, etc.).

While Phase I is primarily focused on the technical feasibility and commercial merit of the tool, the research team seeks to concurrently develop an evaluation design that can robustly assess the impact of the tool along key dimensions that the tool is designed to address:

* Reducing the information processing burden required of patients to navigate the health care system and care plan
* Bridging inefficiencies in the multi-step and multi-stakeholder processes inherent in complex care management and coordination

ELIGIBILITY:
Inclusion Criteria:

* Hepatobiliary surgery patients seeking care at research location
* A sufficient level of comfort with personal computers or smart phone devices

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreas cancer patients and other surgical candidates for procedures including pancreatectomy, whipple procedure.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-26 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Anxiety and Cognitive Burden | Up to 24 weeks
  Patient Health Questionnaire-2 (PHQ-2)
Patient Anxiety and Cognitive Burden | Up to 24 weeks
  Patient Health Questionnaire-9 (PHQ-9)
Time Burden | Through study completion, an average of 6 weeks
  Duration of task completion -- data within the app (time stamps)
Improved information sharing | Through study completion, an average of 8 weeks
  Presence/absence of critical information in app (e.g., imaging)
Improved information sharing | Through study completion, an average of 8 weeks
  Navigator perception via survey feedback

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Downing, Principal Investigator — GMG Arcdata LLC
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States